CLINICAL TRIAL: NCT03158233
Title: Prospective Surveillance and Case Definition Study of Zika Virus Disease and Infection in Adolescents and Adults in Latin America in Preparation for an Efficacy Trial of a Zika Virus Whole Virion, Purified Inactivated Vaccine
Brief Title: Zika Case Definition and Surveillance Study
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: VAG00001
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Zika Virus Disease
Keywords: Zika virus disease
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, surveillance study will assess the operational Zika virus definition for use in future Zika purified inactivated virus (ZIKV) vaccine efficacy trials in order to identify Zika virus disease (ZVD) cases among the study cohort.

DETAILED DESCRIPTION:
This prospective, multicenter, cohort study will conduct active and passive surveillance for ZVD and determine its prevalence and seroconversion incidence in areas of Latin America experiencing Zika epidemic activity. A description of the occurrence of dengue virus and chikungunya virus infections in the cohort may also be provided as differential diagnosis of ZVD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 15 to 40 years on the day of inclusion, currently residing in the site zone, and planning to continue to reside in the site zone for the duration of the study
2. For subjects under the age of majority on the day of inclusion: the assent form has been signed and dated by the subject (if required by local regulations), and the informed consent form has been signed and dated by the parent(s) or legal guardian(s).

For subjects at or over the age of majority on the day of inclusion: the informed consent form has been signed and dated.

3) Subject (and parent/guardian if subject is under the age of majority) able to attend all scheduled visits and to comply with all study procedures 4) In good health, based on medical history and physical examination Exclusion Criteria:

1. Subject is pregnant (as self-reported)
2. Participation in the 4 weeks preceding enrollment, or planned participation during the present study period, in a clinical trial investigating a vaccine, drug, medical device, or a medical procedure
3. Receipt of any dengue or yellow fever vaccine in the 4 weeks preceding the day of enrollment or planned receipt of any dengue or yellow fever vaccine during the study period
4. Receipt of immune globulins, blood or blood-derived products in the past 3 months
5. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
6. History of Zika virus disease, confirmed either clinically, serologically, or virologically
7. Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
8. Current alcohol abuse or drug addiction
9. Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily
10. Identified as an investigator or an employee of the investigator or study center, with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the investigator or employee with direct involvement in the proposed study.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Prospective, multi-center, cohort study in 2400 subjects aged 15 to 40 years at enrollment in 4 countries in Latin America: Colombia, Honduras, Mexico, and Puerto Rico
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with suspected ZVD and virologically confirmed Zika (VCZ) infection in the cohort | Day 0 to Day 365
  Number of suspected ZVD and VCZ infections
Summary of the signs and symptoms accompanying suspected ZVD and VCZ cases in the study participants | Day 0 to Day 365
  Occurrence, intensity, and duration of signs and symptoms of ZVD and VCZ cases

CONTACTS AND LOCATIONS:
Locations (6):
- Colombia (2):
  - Investigational Site, Floridablanca, Santander Department
  - Investigational Site, Cali, Valle del Cauca Department
- Investigational site, Tegucigalpa, Honduras
- Mexico (2):
  - Investigational Site, Acapulco de Juárez, Guerrero
  - Investigational Site, Temixco, Morelos
- Investigational Site, Carolina, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com